CLINICAL TRIAL: NCT03358914
Title: The PsoTeenQOL - Preliminary Reliability and Validity of a Health-related Quality of Life Questionnaire for Adolescents With Psoriasis
Brief Title: The PsoTeenQOL - Preliminary Reliability and Validity
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Herlev and Gentofte Hospital (Other); LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: HRQOL hos unge med psoriasis
Record Dates: First submitted 2017-10-13; First posted 2017-12-02 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Psoriasis
Keywords: psoriasis, adolescents, quality of life, PRO (patient-reported outcome), validation
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Adolescents with psoriasis: No assigned intervention: completion of PsoTeenQOL and other instruments for assessment of psychometric properties and further refinement of the PsoTeenQOL.
  Interventions: Other: No intervention
- Parents of adolescents with psoriasis: No assigned intervention: completion of proxy-version of the PsoTeenQOL for validation purposes
  Interventions: Other: No intervention
- Adolescents without psoriasis: No assigned intervention: completion of non-psoriasis control-version of the PsoTeenQOL for validation purposes
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Completion of surveys

SUMMARY:
This study aims to develop and provide preliminary reliability and validity of a questionnaire to measure Health-related Quality of Life (HRQOL) in adolescents with psoriasis. To the best of our knowledge, this will be the first psoriasis-specific HRQOL instrument for use in adolescent patients. Data will be collected from a Danish population of adolescents with psoriasis (12-17 years), as well as from parents of adolescents with psoriasis, and a group of adolescents without psoriasis.

DETAILED DESCRIPTION:
The present study will examine the psychometric properties of a preliminary 41-item version of the PsoTeenQOL. The preliminary PsoTeenQOL has been developed based on qualitative interviews of adolescents (12-17 years) with psoriasis, their parents, and health professionals working within the field, as well as literature reviews and existing questionnaires. Face and content validity has been established through subsequent cognitive interviews with the target group.

Exploratory factor analysis (EFA) and analysis of differential item functioning (DIF) will be used to further refine the PsoTeenQOL questionnaire by selecting the most appropriate items. In addition, indicators of reliability (internal consistency; test-retest reliability), validity (construct validity, criterion validity; discriminant validity), and responsiveness will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Either a) Subjects with psoriasis, b) Parents of adolescents 12-17 years with psoriasis, or c) Subjects without psoriasis
* Ability to read Danish and complete electronic survey

Exclusion Criteria:

* Inability to read Danish and complete electronic survey

Ages: 12 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: To achieve maximum variation in participant demographic and clinical characteristics, eligible participants with psoriasis plus their parents will be identified through several sites; a) the Danish Psoriasis Association, b) the National Danish Birth Cohort, and c) all five tertiary hospital clinics in Denmark. All adolescents without psoriasis will be recruited from the National Danish Birth Cohort.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Examine the psychometric properties of the PsoTeenQOL | Baseline and up to 3 months after first completion of questionnaire package
  Analyses will include exploratory factor analysis, examination of differential item functioning (DIF) and evaluation of indicators of reliability and validity of the instrument

SECONDARY OUTCOMES:
Indicators of validity | Baseline
  Correlations and comparisons between PsoTeenQOL and similar non-psoriasis-specific instruments (Children's Dermatology Life Quality Index (CDLQI); Pediatric Quality of Life Inventory (PedsQL); WHO-5, proxy- and non-psoriasis control version of the PsoTeenQOL) as well as measures of disease severity (Self-assessed Simplified Psoriasis Index (saSPI), and Psoriasis Area Severity Index (PASI)).
Indicators of reliability | Test-retest: 2 weeks (+/-3 days) after baseline; Responsiveness: 3 months after baseline
  Internal consistencies (Cronbach's alpha), test-retest reliability and responsiveness of the PsoTeenQOL (change scores on the PsoTeenQOL as compared to the CDLQI and disease severity indicators)

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Randa, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No